CLINICAL TRIAL: NCT02510261
Title: A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients With Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Patisiran Clinical Study
Brief Title: The Study of an Investigational Drug, Patisiran (ALN-TTR02), for the Treatment of Transthyretin (TTR)-Mediated Amyloidosis in Participants Who Have Already Been Treated With ALN-TTR02 (Patisiran)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTR02-006; 2014-003877-40 (EudraCT Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-29 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Amyloidosis
Keywords: RNAi therapeutic; FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial | interventions — patisiran

STUDY DESIGN:
Intervention Model Description: All the participants received only patisiran but divided into 3 arm groups based on administration in the parent study (placebo or patisiran in 003 [NCT01961921] or 004 [NCT01960348] studies).
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prior Placebo Group of Study 004 (Experimental): Participants who received placebo and completed parent study ALN-TTR02-004 (NCT01960348) were enrolled to receive 0.3 milligrams per kilogram (mg/kg) patisiran intravenously (IV) once every 3 weeks (Q3W) up to 65.5 months.
  Interventions: Drug: Patisiran
- Prior Patisiran Group of Study 004 (Experimental): Participants who received patisiran and completed parent study ALN-TTR02-004 (NCT01960348) were enrolled to receive 0.3 mg/kg patisiran IV Q3W up to 66.9 months.
  Interventions: Drug: Patisiran
- Prior Patisiran Group of Study 003 (Experimental): Participants who received patisiran and completed parent study ALN-TTR02-003 (NCT01961921) were enrolled to receive 0.3 mg/kg patisiran IV Q3W up to 61.4 months.
  Interventions: Drug: Patisiran

INTERVENTIONS:
Drug: Patisiran — Patisiran was administered IV.
  Other Names: ALN-TTR02

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term dosing with ALN-TTR02 (patisiran) in participants with transthyretin (TTR) mediated amyloidosis (ATTR).

ELIGIBILITY:
Inclusion Criteria:

* Have completed a patisiran study (i.e., completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
* Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

Exclusion Criteria:

* Any new or uncontrolled condition that could make the participant unsuitable for participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (54):
- United States (13):
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Joplin, Missouri
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Cooperstown, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Columbus, Ohio
- Clinical Trial Site, Buenos Aires, Argentina
- Clinical Trial Site, Westmead, Australia
- Brazil (2):
  - Clinical Trial Site, Rio de Janeiro
  - Clinical Trial Site, São Paulo
- Clinical Trial Site, Sofia, Bulgaria
- Clinical Trial Site, Vancouver, British Columbia, Canada
- Clinical Trial Site, Nicosia, Cyprus
- France (6):
  - Clinical Trial Site, Fort de France, Martinique
  - Clinical Trial Site, Saint-Pierre, Reunion Island
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Marseille
- Germany (3):
  - Clinical Trial Site, Cologne
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Münster
- Italy (3):
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Rome
  - Clinical Trial Site, Sicily
- Japan (8):
  - Clinical Trial Site, Ehime
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Hiroshima
  - Clinical Trial Site, Kumamoto
  - Clinical Trial Site, Nagano
  - Clinical Trial Site, Okawasuji
  - Clinical Trial Site, Ono
  - Clinical Trial Site, Ōita
- Clinical Trial Site, Kuala Lumpur, Malaysia
- Clinical Trial Site, Tlalpan, Mexico
- Clinical Trial Site, Groningen, Netherlands
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Clinical Trial Site, Seoul, South Korea
- Spain (4):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Huelva
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Palma de Mallorca
- Clinical Trial Site, Umeå, Sweden
- Clinical Trial Site, Taipei, Taiwan
- Clinical Trial Site, Istanbul, Turkey (Türkiye)
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams D, Wixner J, Polydefkis M, Berk JL, Conceicao IM, Dispenzieri A, Peltier A, Ueda M, Bender S, Capocelli K, Jay PY, Yureneva E, Obici L; patisiran Global OLE study group. Five-Year Results With Patisiran for Hereditary Transthyretin Amyloidosis With Polyneuropathy: A Randomized Clinical Trial With Open-Label Extension. JAMA Neurol. 2025 Mar 1;82(3):228-236. doi: 10.1001/jamaneurol.2024.4631. PMID 39804640
- [Derived] Lin KP, Yang CC, Lee YC, Lee MJ, Vest J, Sweetser MT, White MT, Badri P, Hsieh ST, Chao CC. Patisiran, an RNAi therapeutic for hereditary transthyretin-mediated amyloidosis: Sub-analysis in Taiwanese patients from the APOLLO study. J Formos Med Assoc. 2024 Sep;123(9):975-984. doi: 10.1016/j.jfma.2024.03.008. Epub 2024 Mar 27. PMID 38548524
- [Derived] Adams D, Polydefkis M, Gonzalez-Duarte A, Wixner J, Kristen AV, Schmidt HH, Berk JL, Losada Lopez IA, Dispenzieri A, Quan D, Conceicao IM, Slama MS, Gillmore JD, Kyriakides T, Ajroud-Driss S, Waddington-Cruz M, Mezei MM, Plante-Bordeneuve V, Attarian S, Mauricio E, Brannagan TH 3rd, Ueda M, Aldinc E, Wang JJ, White MT, Vest J, Berber E, Sweetser MT, Coelho T; patisiran Global OLE study group. Long-term safety and efficacy of patisiran for hereditary transthyretin-mediated amyloidosis with polyneuropathy: 12-month results of an open-label extension study. Lancet Neurol. 2021 Jan;20(1):49-59. doi: 10.1016/S1474-4422(20)30368-9. Epub 2020 Nov 16. PMID 33212063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigational sites in Asia, Europe, Canada, the United Kingdom, and the United States from 16 July 2015 to 23 November 2022.
Pre-assignment Details: A total of 211 participants who completed either ALN-TTR02-003 (NCT01961921) or ALN-TTR02-004 (NCT01960348) studies were enrolled into the study to receive at least 1 dose of patisiran.
Period: Overall Study
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Started | 49 | 137 | 25
Full Analysis Set (Full analysis set included all participants who were enrolled in this study.) | 49 | 137 | 25
Safety Analysis Set (Safety analysis set included all the enrolled participants who received at least 1 dose of patisiran in this study.) | 49 | 137 | 25
Pharmacodynamic (PD) Analysis Set (PD analysis set included all participants who received at least 1 dose of patisiran in this study and have had both baseline and at least 1 post-baseline PD assessment (either transthyretin [TTR] or vitamin A).) | 40 | 128 | 24
Completed | 21 | 95 | 22
Not Completed | 28 | 42 | 3
Not completed — Adverse Event | 5 | 8 | 0
Not completed — Physician Decision | 1 | 5 | 0
Not completed — Death | 19 | 19 | 0
Not completed — Withdrawal by Subject | 3 | 10 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were enrolled in this study.
Groups:
- Prior Placebo Group of Study 004: Participants who received placebo and completed parent study ALN-TTR02-004 (NCT01960348) were enrolled to receive 0.3 mg/kg patisiran IV Q3W up to 65.5 months.
- Total: Total of all reporting groups
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003 | Total
Number analyzed (Participants) | 49 | 137 | 25 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.02) | 61.0 (12.10) | 58.5 (15.09) | 61.3 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 35 | 8 | 55
  Male | 37 | 102 | 17 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 2 | 27
  Not Hispanic or Latino | 39 | 121 | 23 | 183
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 14 | 23 | 0 | 37
  Race: Black/African or African American | 0 | 4 | 0 | 4
  Race: White/Caucasian | 34 | 107 | 25 | 166
  Race: Other | 0 | 2 | 0 | 2
  Race: More than One Race | 0 | 1 | 0 | 1
  Race: Missing | 1 | 0 | 0 | 1
Serum Transthyretin (TTR) Level [Mean (Standard Deviation); unit: mg/L] — Population: 'Number analyzed' indicates the number of participants with data available for analysis of the specified measure.
  mg/L
    number analyzed (Participants) | 40 | 128 | 24 | 192
    (all) | 185.689 (56.2895) | 53.010 (43.1782) | 76.905 (47.9088) | 83.639 (70.5576)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Study Discontinuation
Description: AE is any untoward medical occurrence in a participant or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Time Frame: First dose up to 28 days after last dose of study drug (approximately 5.6 years)
Population: Safety analysis set included all the enrolled participants who received at least 1 dose of patisiran in this study. Percentages are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
percentage of participants | 49.0 | 16.8 | 0.0

2. Secondary Outcome: Change From Baseline in the Total Neuropathy Impairment Score (NIS) at Year 5
Description: The NIS assessment is a 244-point composite measure of neurologic impairment which includes a physical exam of lower limbs, upper limbs, and cranial nerves to assess the components: motor strength/weakness (NIS-W), reflexes (NIS-R), and sensation (NIS-S). NIS total score is obtained by combining all the component scores, ranging from 0 to 244. Higher scores represent a greater severity of disease. A positive change from baseline indicates the worsening of neuropathy.
Time Frame: Baseline, Year 5
Population: Full analysis set included all participants who were enrolled in this study. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 81.47 (41.674) | 62.26 (37.875) | 35.48 (28.686)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 92 | 22
  Change From Baseline at Year 5 | 11.45 (16.566) | 10.72 (13.654) | 11.18 (17.554)

3. Secondary Outcome: Change From Baseline in the Total Modified NIS (mNIS +7) Composite Score At Year 3
Description: The mNIS+7 is a composite measure of neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs, and cranial nerves to assess motor strength/weakness (192 points), reflexes (20 points), electrophysiologic measurement of small and large nerve fiber function (10 points), sensory testing (80 points), and postural blood pressure (2 points). The total mNIS+7 composite score is obtained by combining all the component scores, ranging from 0 (no impairment) to 304 (maximum impairment). A negative change from baseline indicates an improvement in neuropathy.
Time Frame: Baseline, Year 3
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 101.07 (43.774) | 74.72 (42.584) | 45.66 (31.640)
  Change From Baseline at Year 3: number analyzed (Participants) | 27 | 105 | 25
  Change From Baseline at Year 3 | -6.69 (3.389) | 8.07 (1.874) | 5.46 (2.450)

4. Secondary Outcome: Change From Baseline in the NIS+7 Total Score at Week 52
Description: The NIS+7 provides additional, objective measures of nerve fibre function and autonomic nerve function in participants with diabetic neuropathy. The NIS+7 includes the full NIS, sum of 5 nerve conduction studies (NCS) (Sural sensory nerve action potential [SNAP], tibial motor nerve distal latency, peroneal compound motor action potential [CMAP], motor nerve conduction velocity, motor nerve distal latency), vibration detection threshold, and pulse rate response to deep breathing. The total NIS+7 score is obtained by combining all the component scores, ranging from 0 (no impairment) to 270 points (maximum impairment). A positive change from baseline indicates worsening.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 98.42 (42.281) | 78.74 (39.417) | 49.66 (31.319)
  Change From Baseline at Week 52: number analyzed (Participants) | 38 | 126 | 25
  Change From Baseline at Week 52 | 1.44 (2.061) | 1.49 (0.894) | 3.23 (2.616)

5. Secondary Outcome: Change From Baseline in the Norfolk Quality of Life-Diabetic Neuropathy (QoL-DN) Questionnaire Total Score at Year 5
Description: The Norfolk QoL-DN questionnaire is a standardized 47-item patient-reported outcomes measure, sensitive to the perception of the effects of diabetic neuropathy by the participant. The scores range from -4 (best possible QOL) to 136 (worst possible QOL). A negative change from baseline represents improved QOL.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline: number analyzed (Participants) | 49 | 137 | 1
  Baseline | 72.7 (28.10) | 54.5 (30.87) | 34.0 (NA) — Standard deviation (SD) cannot be estimated for one participant.
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 94 | 1
  Change From Baseline at Year 5 | 3.3 (13.91) | 4.5 (17.19) | -18.0 (NA) — Standard deviation (SD) cannot be estimated for one participant.

6. Secondary Outcome: Change From Baseline in the EuroQOL-5 Dimensions-5 Levels (EQ-5D-5L) Index Score at Year 5
Description: The EQ-5D-5L is a patient-reported measure of QoL based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The overall score is rated on a scale from 0 (worst) to 1 (no impairment). Higher scores indicate a higher QoL. A negative change from baseline indicates worsening of QoL.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 0.4614 (0.03347) | 0.6444 (0.01856) | 0.7663 (0.03336)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 94 | 21
  Change From Baseline at Year 5 | 0.0361 (0.04017) | -0.0548 (0.01767) | -0.0166 (0.02363)

7. Secondary Outcome: Change From Baseline in the EuroQoL Visual Analogue Scale (EQ-VAS) Score at Year 5
Description: EQ-VAS measures the participant's self-rated health on a vertical scale evaluated on a scale of 0 ("worst health you can imagine") to 100 ("best health you can imagine"). Higher scores indicate a higher QOL. A negative change from baseline indicates worsening of QoL.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 46.0 (2.86) | 57.8 (1.82) | 69.1 (4.20)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 94 | 22
  Change From Baseline at Year 5 | 9.3 (5.03) | -1.5 (1.43) | 1.5 (2.99)

8. Secondary Outcome: Change From Baseline in the Composite Autonomic Symptom Score (COMPASS 31) Total Score at Week 52
Description: COMPASS 31 questionnaire measures autonomic symptoms in participants with neuropathy. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor). COMPASS 31 is measured on a scale from 0 to 100, with 100 representing maximum impairment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 33.92 (18.185) | 25.37 (17.010) | 15.93 (15.116)
  Change From Baseline at Week 52: number analyzed (Participants) | 38 | 126 | 25
  Change From Baseline at Week 52 | -3.70 (12.957) | 0.37 (12.041) | -1.24 (7.975)

9. Secondary Outcome: Change From Baseline in the Modified Body Mass Index (mBMI) at Year 5
Description: Nutritional status of participants was evaluated using the mBMI, calculated as BMI (kilograms per square meter [kg/m^2]) multiplied by the concentration of serum albumin (grams per liter [g/L]). A positive change from baseline indicates improvement in nutritional status.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg.g/m^2.L
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
kg.g/m^2.L
  Baseline | 881.8 (219.10) | 970.7 (218.40) | 1002.3 (173.80)
  Change From Baseline at Year 5: number analyzed (Participants) | 20 | 84 | 22
  Change From Baseline at Year 5 | 74.0 (146.85) | 31.6 (119.28) | 77.8 (91.36)

10. Secondary Outcome: Change From Baseline in the Rasch-built Overall Disability Scale (R-ODS) at Year 5
Description: The R-ODS is a 24-item patient-reported questionnaire that specifically captures activity and social participation limitations. It measures the level of disability on a scale of 0 (worst) to 48 (best, no limitations), higher score indicates a better outcome. A negative change from baseline indicates worsening of disability.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 20.3 (12.74) | 29.7 (12.56) | 36.7 (10.29)
  Change From Baseline at Year 5: number analyzed (Participants) | 20 | 93 | 22
  Change From Baseline at Year 5 | -2.9 (5.25) | -4.1 (6.78) | -2.7 (3.60)

11. Secondary Outcome: Change From Baseline in the NIS+7 Component: NIS-Weakness (NIS-W) Score at Year 5
Description: The NIS+7 provides additional, objective measures of nerve fiber function and autonomic nerve function in participants with diabetic neuropathy. The NIS+7 includes the full NIS (NIS-W, NIS-R, NIS-S), sum of 5 nerve conduction studies (NCS) (Sural SNAP, tibial motor nerve distal latency, peroneal CMAP, motor nerve conduction velocity, motor nerve distal latency), vibration detection threshold, and pulse rate response to deep breathing. NIS-W is a measure of motor strength, comprised of cranial nerve and both upper and lower limb motor assessments. The score ranges from 0 to 192. A higher score indicates greater severity of disease.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
score on a scale
  Baseline | 47.01 (31.323) | 33.26 (27.434) | 15.02 (17.988)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 92 | 22
  Change From Baseline at Year 5 | 9.10 (13.297) | 7.37 (11.707) | 6.97 (13.235)

12. Secondary Outcome: Change From Baseline in the 10-meter Walk Test (10-MWT) Speed at Year 5
Description: 10-MWT is a measure of ambulatory ability and walk speed. It measures the speed (in meters per second [m/s]) of a participant to walk 10 meters. A negative change from baseline represents decreased ambulatory ability.
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
m/s
  Baseline | 0.538 (0.0553) | 0.851 (0.0422) | 1.262 (0.0826)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 92 | 22
  Change From Baseline at Year 5 | 0.011 (0.0339) | -0.050 (0.0542) | -0.121 (0.0487)

13. Secondary Outcome: Change From Baseline in the Hand Grip Strength at Week 52
Description: Hand grip strength was measured by dynamometer. Grip strength in the dominant arm is a measure of motor function, with a higher grip strength indicating better motor function. The mean change from baseline in the hand grip strength was reported.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: kg
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
kg
  Baseline | 10.23 (1.293) | 18.03 (1.081) | 27.86 (2.626)
  Change From Baseline at Week 52: number analyzed (Participants) | 38 | 125 | 25
  Change From Baseline at Week 52 | 0.14 (0.461) | -0.34 (0.615) | -0.28 (0.807)

14. Secondary Outcome: Number of Participants With Change From Baseline in the Polyneuropathy Disability (PND) Stage
Description: PND measures changes in the ambulatory ability including the need of walking aids on the following stages: 0 (no symptoms), I (sensory disturbances but preserved walking capability), II (impaired walking capability but ability to walk without a stick or crutches), IIIA (walking with help of 1 stick/crutch), IIIB (with help of 2 sticks/crutches), and IV (confined to wheelchair or bedridden). Lower scores indicate greater ambulatory function. The number of participants with change in the stage from baseline was reported as: Improved or worsened.
Time Frame: Baseline, Year 5
Population: Full analysis set included all participants who were enrolled in this study. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 21 | 94 | 22
Participants
  Improved | 1 | 9 | 3
  Worsened | 8 | 35 | 5

15. Secondary Outcome: Number of Participants With Change From Baseline in the Familial Amyloidotic Polyneuropathy (FAP) Stage
Description: FAP measures changes in the ambulatory ability including the need of walking aids on the following stages: 0 (no symptoms), I (unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs), II (assistance with ambulation required; moderate impairment of the lower limbs, upper limbs, and trunk), and III (wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs). Lower scores indicate greater ambulatory function. The number of participants with change in the stage from baseline was reported as: Improved or worsened.
Time Frame: Baseline, Year 5
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 21 | 93 | 22
Participants
  Improved | 0 | 3 | 1
  Worsened | 5 | 13 | 2

16. Secondary Outcome: Number of Participants With Change From Baseline in the New York Heart Association (NYHA) Classification
Description: NYHA classification grades the severity of heart failure symptoms into the following stages: I (no symptoms; ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea), II (symptoms with ordinary physical activity; walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea), III (symptoms with less than ordinary physical activity; walking 1 to 2 blocks on the level and climbing more than 1 flight of stairs in normal conditions causes undue fatigue or dyspnea), IV (symptoms at rest; inability to carry on any physical activity without fatigue or dyspnea). The number of participants with change in the stage from baseline was reported as: Improved or worsened.
Time Frame: Baseline, Year 5
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 20 | 87 | 21
Participants
  Improved | 2 | 13 | 1
  Worsened | 4 | 18 | 4

17. Secondary Outcome: Change From Baseline in the Intraepidermal Nerve Fiber Density (IENFD) at Year 5
Description: IENFD (fibers/millimeter [mm]) is a measure for the pathologic evaluation of sensory and autonomic innervation. It is obtained by tandem 3 mm skin punch biopsies: one set of biopsies taken from the distal thigh and one set from the distal lower leg. An increase in nerve fiber density suggests improvement, while a decrease in nerve fiber density suggests worsening.
Time Frame: Baseline, Year 5
Population: Full analysis set included all participants who were enrolled in this study. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis of the specified parameter at specified timepoint.
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 15 | 61 | 19
fibers/mm
  Epidermal Nerve Fibers, Thigh: Baseline | 4.71 (5.249) | 5.41 (5.291) | 8.99 (10.027)
  Epidermal Nerve, Fibers, Thigh: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 15 | 11
  Epidermal Nerve, Fibers, Thigh: Change From Baseline at Year 5 | 0.28 (2.298) | -2.75 (3.126) | -5.53 (7.998)
  Epidermal Nerve Fibers, Leg: Baseline: number analyzed (Participants) | 13 | 60 | 18
  Epidermal Nerve Fibers, Leg: Baseline | 0.47 (0.843) | 1.70 (3.183) | 3.66 (8.286)
  Epidermal Nerve Fibers, Leg: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 15 | 11
  Epidermal Nerve Fibers, Leg: Change From Baseline at Year 5 | -0.25 (0.495) | -1.31 (1.879) | -3.50 (8.428)

18. Secondary Outcome: Change From Baseline in the Sweat Gland Nerve Fiber Density (SGNFD) at Year 5
Description: SGNFD (meter/cubic millimeter [m/mm^3]) is a measure for the pathologic evaluation of sensory and autonomic innervation. It is obtained by tandem 3 mm skin punch biopsies: one set of biopsies taken from the distal thigh and one set from the distal lower leg. An increase in nerve fiber density suggests improvement, while a decrease in nerve fiber density suggests worsening.
Time Frame: Baseline, Year 5
Population: Full analysis set included all participants who were enrolled in this study. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number of participants analyzed' indicates the number of participants with data available for analysis of the specified parameter at specified timepoint.
Measure: Mean (Standard Deviation); unit: m/mm^3
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 15 | 59 | 19
m/mm^3
  Sweat Gland Nerve Fibers, Thigh: Baseline | 10.82 (6.638) | 9.67 (4.942) | 9.14 (4.802)
  Sweat Gland Nerve Fibers, Thigh: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 14 | 10
  Sweat Gland Nerve Fibers, Thigh: Change From Baseline at Year 5 | -0.56 (2.648) | -2.49 (5.636) | -3.29 (4.323)
  Sweat Gland Nerve Fibers, Leg: Baseline: number analyzed (Participants) | 13 | 59 | 18
  Sweat Gland Nerve Fibers, Leg: Baseline | 2.82 (3.363) | 4.99 (4.274) | 5.93 (4.355)
  Sweat Gland Nerve Fibers, Leg: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 15 | 9
  Sweat Gland Nerve Fibers, Leg: Change From Baseline at Year 5 | 1.43 (2.351) | -2.47 (3.605) | -1.31 (2.867)

19. Secondary Outcome: Change From Baseline in the Dermal Amyloid Burden at Year 5
Description: Dermal Amyloid Burden is a measure for the pathologic evaluation of sensory and autonomic innervation and reported as % congo red stain. It is obtained by tandem 3 mm skin punch biopsies: one set of biopsies taken from the distal thigh and one set from the distal lower leg.
Time Frame: Baseline, Year 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent congo red stain
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 15 | 61 | 18
percent congo red stain
  Amyloid Stain, Thigh: Baseline | 8.163 (10.6544) | 8.205 (10.8725) | 5.908 (7.6646)
  Amyloid Stain, Thigh: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 15 | 10
  Amyloid Stain, Thigh: Change From Baseline at Year 5 | -3.775 (5.3387) | -1.103 (7.5569) | -3.100 (5.7269)
  Amyloid Stain, Leg: Baseline: number analyzed (Participants) | 13 | 60 | 17
  Amyloid Stain, Leg: Baseline | 11.062 (10.4857) | 10.386 (12.3967) | 7.441 (8.5566)
  Amyloid Stain, Leg: Change From Baseline at Year 5: number analyzed (Participants) | 2 | 15 | 10
  Amyloid Stain, Leg: Change From Baseline at Year 5 | -7.475 (5.6922) | -2.793 (6.2309) | -3.935 (6.6372)

20. Secondary Outcome: Change From Baseline in the Cardiac Biomarker: Serum Troponin I at Year 5
Description: Manifestations of cardiac amyloid involvement were assessed through measurement of serum levels of the cardiac biomarker: troponin (micrograms per liter [µg/L]). The troponin I values <0.1 μg/L were imputed to 0.1 thus the actual changes cannot be calculated for values <0.1 μg/L.
Time Frame: Baseline, Year 5
Population: Full analysis set included all participants who were enrolled in this study. 'Number analyzed' indicates the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
µg/L
  Baseline | 0.109 (0.0360) | 0.112 (0.0963) | 0.088 (0.0263)
  Change From Baseline at Year 5: number analyzed (Participants) | 18 | 85 | 22
  Change From Baseline at Year 5 | 0.546 (2.3345) | -0.005 (0.0244) | 0.014 (0.0277)

21. Secondary Outcome: Change From Baseline in the Cardiac Biomarker: N-terminal Prohormone of B-type Natriuretic Peptide (NT-proBNP) at Year 5
Description: Manifestations of cardiac amyloid involvement were assessed through measurement of serum levels of the cardiac biomarker: NT-proBNP (nanograms per liter [ng/L]).
Time Frame: Baseline, Year 5
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
ng/L
  Baseline | 1957.649 (2731.3296) | 1017.217 (1558.7632) | 281.899 (421.9627)
  Change From Baseline at Year 5: number analyzed (Participants) | 19 | 84 | 21
  Change From Baseline at Year 5 | -18.490 (910.2156) | 209.126 (487.2140) | 78.146 (266.1912)

22. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: Average Peak Longitudinal Strain at Year 5
Description: The echocardiogram parameters analyzed included measures of systolic function: Average peak longitudinal strain (percentage [%]).
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 136 | 25
percentage
  Baseline | -15.63 (3.348) | -15.96 (3.283) | -17.72 (4.079)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 87 | 22
  Change From Baseline at Year 5 | 3.43 (3.634) | 2.30 (3.300) | 1.62 (3.082)

23. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: Left Ventricular (LV) Mass at Year 5
Description: The echocardiogram parameters analyzed included measures of cardiac structure: LV mass (grams [g]).
Time Frame: Baseline, Year 5
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
grams
  Baseline | 238.166 (74.0536) | 236.604 (85.8152) | 198.570 (89.1780)
  Change From Baseline at Year 5: number analyzed (Participants) | 20 | 89 | 22
  Change From Baseline at Year 5 | 2.723 (52.1737) | -4.222 (48.2397) | -17.152 (50.9296)

24. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: LV End-diastolic Volume at Year 5
Description: The echocardiogram parameters analyzed included measures of diastolic function: LV end-diastolic volume (milliliters [mL]).
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 136 | 25
mL
  Baseline | 80.591 (26.5862) | 83.616 (25.6990) | 107.818 (34.8418)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 84 | 21
  Change From Baseline at Year 5 | 7.173 (15.9316) | -1.279 (20.0305) | -11.710 (32.1329)

25. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: LV Relative Wall Thickness at Year 5
Description: The echocardiogram parameters analyzed included measures of cardiac structure: LV relative wall thickness (ratio).
Time Frame: Baseline, Year 5
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
ratio
  Baseline | 0.780 (0.1616) | 0.717 (0.1840) | 0.593 (0.1802)
  Change From Baseline at Year 5: number analyzed (Participants) | 20 | 89 | 22
  Change From Baseline at Year 5 | -0.066 (0.1344) | -0.061 (0.1320) | -0.037 (0.0887)

26. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: Mean LV Wall Thickness at Year 5
Description: The echocardiogram parameters analyzed included measures of cardiac structure: Mean LV wall thickness (centimeters [cm]).
Time Frame: Baseline, Year 5
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Prior Placebo Group of Study 004: Participants who received placebo and completed parent study ALN-TTR02-004 (NCT01960348) were enrolled to receive 0.3 mg/kg patisiran IVQ3W up to 65.5 months.
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 137 | 25
cm
  Baseline | 1.538 (0.2776) | 1.463 (0.3210) | 1.249 (0.3321)
  Change From Baseline at Year 5: number analyzed (Participants) | 20 | 89 | 22
  Change From Baseline at Year 5 | -0.035 (0.1782) | -0.041 (0.1874) | -0.042 (0.1794)

27. Secondary Outcome: Change From Baseline in the Echocardiogram Parameter: Cardiac Output at Year 5
Description: The echocardiogram parameters analyzed included measures of systolic function: Cardiac output (liters per minute [L/min]).
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 49 | 136 | 25
L/min
  Baseline | 3.547 (1.0373) | 3.840 (1.1748) | 4.873 (1.6902)
  Change From Baseline at Year 5: number analyzed (Participants) | 21 | 83 | 21
  Change From Baseline at Year 5 | -0.010 (1.1551) | -0.283 (1.1012) | -0.594 (1.5476)

28. Secondary Outcome: Percent Change From Baseline in Serum TTR Levels at Year 5
Description: Serum TTR was assessed using enzyme linked immunosorbent assay (ELISA).
Time Frame: Baseline, Year 5
Population: PD analysis set included all participants who received at least 1 dose of patisiran in this study and have had both baseline and at least 1 post-baseline PD assessment (either TTR or vitamin A). 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
Number analyzed (Participants) | 19 | 80 | 21
percent change | -90.010 (7.4802) | -37.660 (35.2948) | -39.965 (56.5274)

ADVERSE EVENTS:
Time Frame: First dose up to 28 days after last dose of study drug (approximately 5.6 years)
Description: Safety analysis set included all the enrolled participants who received at least 1 dose of patisiran in this study.
Arm/Group | Prior Placebo Group of Study 004 | Prior Patisiran Group of Study 004 | Prior Patisiran Group of Study 003
All-Cause Mortality (participants affected / at risk) | 19/49 | 21/137 | 1/25
Serious Adverse Events (participants affected / at risk) | 39/49 | 82/137 | 12/25
Other Adverse Events (participants affected / at risk) | 47/49 | 135/137 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo Group of Study 004 (N=49) | Prior Patisiran Group of Study 004 (N=137) | Prior Patisiran Group of Study 003 (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 2 | 0
Arrhythmia (Cardiac disorders) | 2 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 6 | 0
Atrial Flutter (Cardiac disorders) | 0 | 4 | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 1 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 3 | 3 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Cardiac Amyloidosis (Cardiac disorders) | 1 | 4 | 0
Cardiac Arrest (Cardiac disorders) | 5 | 0 | 0
Cardiac Failure (Cardiac disorders) | 2 | 4 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 2 | 0
Cardiac Flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 1 | 0
Conduction Disorder (Cardiac disorders) | 0 | 3 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0 | 0
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Familial Amyloidosis (Congenital, familial and genetic disorders) | 1 | 2 | 0
Hereditary Neuropathic Amyloidosis (Congenital, familial and genetic disorders) | 1 | 1 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 2 | 0
Corneal Perforation (Eye disorders) | 0 | 1 | 0
Deposit Eye (Eye disorders) | 2 | 0 | 0
Eye Haemorrhage (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Retinal Artery Occlusion (Eye disorders) | 1 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 2 | 0
Retinal Ischaemia (Eye disorders) | 0 | 1 | 0
Rhegmatogenous Retinal Detachment (Eye disorders) | 0 | 1 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 2 | 0
Vitreous Opacities (Eye disorders) | 0 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Faeces Pale (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Asthenia (General disorders) | 2 | 2 | 0
Chest Discomfort (General disorders) | 0 | 0 | 1
Extravasation (General disorders) | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 1 | 0
Generalised Oedema (General disorders) | 0 | 1 | 0
Implant site injury (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Polyp (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Sudden Cardiac Death (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 2 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0
COVID-19 Pneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 5 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Infusion Site Cellulitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Parotitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 5 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 1 | 0
Septic Shock (Infections and infestations) | 2 | 2 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 4 | 0
Urosepsis (Infections and infestations) | 1 | 2 | 0
Vascular Device Infection (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured Sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stoma Site Extravasation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Intraocular Pressure Increased (Investigations) | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Amyloid Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ocular Surface Squamous Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 | 2 | 0
Basal Ganglia Infarction (Nervous system disorders) | 0 | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Hypoxic-ischaemic Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Psychomotor Skills Impaired (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 4 | 1
Device Capturing Issue (Product Issues) | 0 | 1 | 0
Device Physical Property Issue (Product Issues) | 0 | 1 | 0
Device Power Source Issue (Product Issues) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Conversion Disorder (Psychiatric disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 1
Calculus Bladder (Renal and urinary disorders) | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1 | 0
End Stage Renal Disease (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Neurogenic Bladder (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Disability (Social circumstances) | 0 | 1 | 0
Rehabilitation Therapy (Social circumstances) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 2 | 0 | 0
Neurogenic Shock (Vascular disorders) | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Poor Peripheral Circulation (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Shock Haemorrhagic (Vascular disorders) | 2 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo Group of Study 004 (N=49) | Prior Patisiran Group of Study 004 (N=137) | Prior Patisiran Group of Study 003 (N=25)
Anaemia (Blood and lymphatic system disorders) | 7 | 10 | 2
Arrhythmia (Cardiac disorders) | 3 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 14 | 0
Atrial Flutter (Cardiac disorders) | 1 | 2 | 2
Cardiac Failure (Cardiac disorders) | 4 | 3 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 15 | 4
Vertigo Positional (Ear and labyrinth disorders) | 0 | 3 | 2
Cataract (Eye disorders) | 5 | 14 | 5
Conjunctival Haemorrhage (Eye disorders) | 5 | 4 | 1
Visual Impairment (Eye disorders) | 1 | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 10 | 1
Abdominal Pain Upper (Eye disorders) | 6 | 4 | 1
Constipation (Gastrointestinal disorders) | 9 | 19 | 3
Dental Caries (Gastrointestinal disorders) | 1 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 22 | 35 | 3
Dry Mouth (Gastrointestinal disorders) | 4 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 2 | 0
Flatulence (Gastrointestinal disorders) | 3 | 3 | 0
Gastritis (Gastrointestinal disorders) | 4 | 7 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 5 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 7 | 0
Nausea (Gastrointestinal disorders) | 10 | 22 | 3
Toothache (Gastrointestinal disorders) | 4 | 8 | 2
Vomiting (Gastrointestinal disorders) | 5 | 14 | 3
Asthenia (General disorders) | 5 | 10 | 1
Fatigue (General disorders) | 1 | 6 | 2
Gait Disturbance (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 1 | 4 | 2
Oedema Peripheral (General disorders) | 15 | 35 | 6
Peripheral Swelling (General disorders) | 4 | 8 | 0
Pyrexia (General disorders) | 5 | 18 | 3
Infusion Related Reaction (Immune system disorders) | 13 | 17 | 4
Bronchitis (Infections and infestations) | 1 | 7 | 1
COVID-19 (Infections and infestations) | 3 | 13 | 0
Cellulitis (Infections and infestations) | 2 | 9 | 0
Conjunctivitis (Infections and infestations) | 4 | 7 | 0
Erysipelas (Infections and infestations) | 1 | 5 | 3
Eye infection (Infections and infestations) | 3 | 0 | 0
Fungal skin infection (Infections and infestations) | 4 | 4 | 2
Gastroenteritis (Infections and infestations) | 2 | 8 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 1 | 3
Influenza (Infections and infestations) | 6 | 18 | 4
Localised Infection (Infections and infestations) | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 9 | 28 | 8
Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 3
Rhinitis (Infections and infestations) | 1 | 9 | 1
Sinusitis (Infections and infestations) | 0 | 5 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 21 | 1
Urinary Tract Infection (Infections and infestations) | 16 | 28 | 5
Wound Infection (Infections and infestations) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 8 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 33 | 5
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 10 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 10 | 1
Limb Injury (Injury, poisoning and procedural complications) | 6 | 14 | 6
Post-traumatic Pain (Injury, poisoning and procedural complications) | 3 | 5 | 2
Skin Abrasion (Injury, poisoning and procedural complications) | 3 | 9 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 6 | 11 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 2 | 9 | 2
N-terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 3 | 3 | 0
Weight Decreased (Investigations) | 4 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 8 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 7 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 15 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 21 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 13 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 12 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 29 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 11 | 21 | 1
Headache (Nervous system disorders) | 11 | 19 | 1
Neuralgia (Nervous system disorders) | 2 | 12 | 2
Paraesthesia (Nervous system disorders) | 0 | 4 | 2
Sciatica (Nervous system disorders) | 3 | 8 | 1
Somnolence (Nervous system disorders) | 4 | 7 | 0
Syncope (Nervous system disorders) | 6 | 11 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 2
Depression (Psychiatric disorders) | 4 | 8 | 2
Insomnia (Psychiatric disorders) | 7 | 11 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 2 | 1
Dysuria (Renal and urinary disorders) | 3 | 8 | 1
Haematuria (Renal and urinary disorders) | 3 | 9 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 2
Urinary Retention (Renal and urinary disorders) | 3 | 3 | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 4 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 20 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 4 | 7 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 12 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 5 | 7 | 3
Flushing (Vascular disorders) | 4 | 5 | 5
Hypertension (Vascular disorders) | 2 | 16 | 2
Hypotension (Vascular disorders) | 3 | 16 | 0
Orthostatic Hypotension (Vascular disorders) | 3 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT02510261/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT02510261/SAP_001.pdf